CLINICAL TRIAL: NCT00221650
Title: Efficacy and Safety of Peginterferon alfa2a and Ribavirin for the Second Line Treatment of Chronic Hepatitis C in HIV Infected Patients Previously Non Responders to a First Anti-HCV Treatment
Brief Title: Treatment of Chronic Hepatitis C With PEG Interferon alfa2a and Ribavirin in HIV-Infected Patients
Acronym: ROCO2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Hoffmann-La Roche (Industry); Ministry of Health, France (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9232-01; 2000-023
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: HIV Infections; Hepatitis C, Chronic; Treatment Failure
Keywords: Hepatitis C, Chronic; HCV infection; HIV infection; Treatment Failure; PEG interferon; Interferons/therapeutic use; Interferon Alfa-2a/adverse effects; Ribavirin/therapeutic use; Ribavirin/adverse effects; Drug Therapy, Combination; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections; Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Peginterferon alfa2a
Drug: Ribavirin

SUMMARY:
Combination of PEG interferon and ribavirin is the standard treatment of chronic hepatitis C. Efficacy of this treatment has never been evaluated in HCV-HIV infected patients, who have previously been treated with a first line anti-HCV treatment. The purpose of the study is to evaluate the combination PEG interferon alfa2a-ribavirin in HIV-infected patients with chronic hepatitis C pretreated with interferon alone or interferon combined with ribavirin. The patients receive a dose of 180 µg of PEGASYS once a week and 800 to 1200 mg/day of ribavirin (according to weight) for 48 weeks. Primary outcome of the study is a sustained virological response, defined as an undetectable HCV RNA level 24 weeks after the end of anti-HCV treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C : Detectable HCV RNA, Previously treated with interferon or interferon combined with ribavirin, Elevated ALT level
* HIV infection (CD4>250/µL, HIV RNA<10 000 copies/ml) treated or not with antiretroviral therapy
* Signed informed consent

Exclusion Criteria:

* Chronic hepatitis B
* Alcohol consumption>40g/day
* Evidence of decompensated liver disease
* Hepatocellular carcinoma
* Other relevant disorders: organ transplantation, psychiatric or cardiovascular disease, poorly controlled diabetes, seizure disorders, hemoglobinopathy, autoimmune disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2002-04; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a sustained virological response, defined as an undetectable HCV RNA level | 24 weeks after the end of anti-HCV treatment

SECONDARY OUTCOMES:
Proportion of patients with a virological response | at weeks 24 and 48
Safety of treatment
Influence of anti-HCV treatment on CD4 count and HIV RNA
Proportion of patients with histological response 24 weeks after the end of anti-HCV treatment

CONTACTS AND LOCATIONS:
Overall Officials: Didier Neau, MD-PhD, Principal Investigator — Hôpital Pellegrin, 33076 Bordeaux Cedex, France; Genevieve Chene, Pr, Study Chair — University Hospital, Bordeaux
Locations (1):
- Hôpital Pellegrin, Federation des Maladies Infectieuses, Pr RAGNAUD, Bordeaux, France

REFERENCES:
- [Background] Thiebaut R, Guedj J, Jacqmin-Gadda H, Chene G, Trimoulet P, Neau D, Commenges D. Estimation of dynamical model parameters taking into account undetectable marker values. BMC Med Res Methodol. 2006 Aug 1;6:38. doi: 10.1186/1471-2288-6-38. PMID 16879756